CLINICAL TRIAL: NCT00552396
Title: An Open-label, Dose-escalation Safety and Tolerability Trial Assessing Multiple Dose Administrations of Anti-KIR (1-7F9) Human Monoclonal Antibody in Subjects With Multiple Myeloma
Brief Title: An Open-label, Dose-escalation Safety and Tolerability Trial Assessing Anti-KIR (1-7F9) in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH2101-103
Record Dates: First submitted 2007-05-21; First posted 2007-11-01 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Anti-KIR (1-7F9)
MeSH Terms: conditions — Multiple Myeloma | interventions — IPH-2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Anti-KIR (1-7F9) — human monoclonal antibody

SUMMARY:
Development of new treatments for diseases such as multiple myeloma is a focus for research. The research being conducted is on treatment called Anti-KIR (1-7F9), which activates the body's own cells to kill tumor cells. This is different from many other treatments where chemicals are given to kill tumor cells. The purpose of the study is to determine a safe dose of Anti-KIR (1-7F9) to administer in humans and to gain information about its effectiveness in the treatment of multiple myeloma.

DETAILED DESCRIPTION:
Trial Design:

The trial is an open-label, dose-escalation trial to determine the safety and tolerability of Anti-KIR (1-7F9) in subjects with relapsed or refractory multiple myeloma (RRMM). A 3+3 design will be employed for the first dosing cycle at each dose level. The 7 planned dose levels are 0.0003 mg/kg, 0.003 mg/kg, 0.015 mg/kg, 0.075 mg/kg, 0.3 mg/kg, 1.0 mg/kg and 3.0 mg/kg. The subjects will receive up to a total of 4 administrations of Anti-KIR (1-7F9) with a dosing interval between each administration of 4 weeks. Safety, toxicity, PK (pharmacokinetic) and PD (pharmacodynamic) obtained in the first 4 weeks after dosing per group will be the basis for dose-escalation decisions. There will be follow-up visits every week the one month after the first administration and every two weeks following the second, third and fourth administrations. After the last administration there will be follow-up visits every month until KIR occupancy is no longer detected.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
2. Bone marrow plasmacytosis > 10% (as determined by bone marrow aspirate) or plasmacytoma
3. Relapse or progression after at least one prior systemic treatment regimen for Multiple Myeloma (MM) as evidenced by ≥ 25% increase in the M-protein as compared to the best response from the previous treatment regimen.

3a. One prior therapy for multiple myeloma, Measurable disease, as defined by persistent presence of serum and/or urine monoclonal protein or abnormal serum free light chain ratio following the prior treatment.

a. Only for the last seven patients enrolled into the cohort 7 or Maximal Tolerated Dose (MTD).

4. Full recovery from acute toxicities of prior anti-MM therapies. 5. Peripheral blood (Natural Killer) NK cells (Absolute CD16, 56)≥ 0.05 x 109/L (50/mm3) 6. Detectable binding of Anti-KIR (1-7F9) to subject NK cells 7. Age ≥ 18 years 8. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2 9. Clinical laboratory values at screening:

* serum creatinine < grade 2 toxicity i.e. 1.5x upper limit of institutional normal value
* total bilirubin < 1.5x upper limit of institutional normal value
* Aspartate aminotransferase (AST) < or = 3x upper limit of institutional normal value
* Absolute Neutrophil Count (ANC) >1.2 x109/L
* Platelets >70x109/L

Exclusion Criteria:

1. Known or suspected allergy to trial product or related products
2. Previous participation in this trial (dosed)
3. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (appropriate methods include abstinence and the following methods: diaphragm, condom (by the partner), intrauterine device, sponge, spermicide or oral contraceptives)
4. Male subjects who are sexually active and have not been surgically sterilized must be informed that they must either use a condom during intercourse, ensure that their partners practices contraception, or they must refrain from sexual intercourse during the study and until 1 month after completion of the trial.
5. Use of an investigational agent within 30 days of the first dose of study drug (or five half-lives of any antibody).
6. Current treatment with any other anti-MM therapy excluding prophylactic bisphosphonates.
7. Radiotherapy against bone lesions within 4 weeks or visceral lesions within 8 weeks of Screening.
8. Thalidomide or bortezomib treatment within 14 days of Screening.
9. Cytotoxic chemotherapy (excluding thalidomide or bortezomib) or corticosteroid treatment within 28 days of Screening.
10. Subjects with non-secretory multiple myeloma
11. Subjects on dialysis
12. Use of myeloid growth factor within 28 days of screening
13. G-CSF treatment within 28 days of screening
14. Active autoimmune disease
15. Active infectious disease (e.g. HIV, chronic hepatitis, etc.) as judged by the investigator.
16. New York Heart Association (NYHA) class III-IV heart failure
17. Severe neurological / psychiatric disorder as judged by the investigator
18. Clinical evidence of an active second malignancy, with the exception of basal cell carcinoma or in situ carcinoma of cervix.
19. Subjects with a history of allogenic transplantation.
20. Subject who have undergone autologous transplantation within the last 3 months.
21. Mental incapacity or inadequate understanding of English.
22. Any serious medical condition that in the opinion of the investigator, disqualifies the subject for inclusion in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — Indiana University; Don Benson, Jr., MD, PhD, Principal Investigator — Division of Haematology/Oncology - Ohio State University; Swaminathan Padmanabhan, MD, Principal Investigator — CTRC Institute for Drug Development - University of Texas at San Antonio; Sundar Jagannath, MD, Principal Investigator — Mount Sinai Hospital, New York
Locations (4):
- United States (4):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Mont Sinai Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Cancer Therapy Research Center at UTHSCSA, San Antonio, Texas

REFERENCES:
- [Derived] Benson DM Jr, Hofmeister CC, Padmanabhan S, Suvannasankha A, Jagannath S, Abonour R, Bakan C, Andre P, Efebera Y, Tiollier J, Caligiuri MA, Farag SS. A phase 1 trial of the anti-KIR antibody IPH2101 in patients with relapsed/refractory multiple myeloma. Blood. 2012 Nov 22;120(22):4324-33. doi: 10.1182/blood-2012-06-438028. Epub 2012 Oct 1. PMID 23033266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 subjects were enrolled and 21 subjects were screen failures
Groups:
- 0.0003 mg/kg: 3+3 design was employed for the first dosing cycle at each dose level. The 7 dose levels were 0.0003 mg/kg, 0.003 mg/kg, 0.015 mg/kg, 0.075 mg/kg, 0.3 mg/kg, 1.0 mg/kg, and 3.0 mg/kg. The subjects received up to a total of 4 administrations of Anti-KIR (1-7F9) with a dosing interval between each administration of 4 weeks.
Period: Overall Study
Arm/Group | 0.0003 mg/kg | 0.003 mg/kg | 0.015 mg/kg | 0.075 mg/kg | 0.3 mg/kg | 1 mg/kg | 3 mg/kg
Started | 4 | 3 | 3 | 6 | 3 | 3 | 10
Completed | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 3 | 3 | 3 | 6 | 3 | 3 | 9
Not completed — protocol withdrawal criteria | 3 | 3 | 3 | 6 | 3 | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.0003 mg/kg | 0.003 mg/kg | 0.015 mg/kg | 0.075 mg/kg | 0.3 mg/kg | 1 mg/kg | 3 mg/kg | Total
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 3 | 10 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 3 | 1 | 2 | 7 | 21
  >=65 years | 1 | 0 | 1 | 3 | 2 | 1 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (4.03) | 49.7 (2.52) | 66 (11.53) | 64 (5.51) | 62.7 (11.02) | 60.3 (7.57) | 60.6 (18.68) | 61.1 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3 | 1 | 2 | 4 | 13
  Male | 3 | 2 | 2 | 3 | 2 | 1 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 6 | 3 | 3 | 10 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of IPH2101 as Determined by Number of Participants With Dose-Limiting Toxicities (DLTs) Related to IPH2101 Treatment
Description: The maximum tolerated dose (MTD) is the highest dose level below the maximum administered dose (MAD) where none or 1 out of 6 subjects have a DLT.
Time Frame: From start of the treatment to end of study
Population: All treated participants who received at least one dose of the study drug and were evaluable for DLT
Measure: Number; unit: Number of participants with DLT
Groups:
- IPH2101 0.0003 mg/kg: Participants were administered an IV dose of 0.0003 mg/kg IPH2101 every 4 weeks for 4 cycles. Initially, 3 participants were treated at one dose level. If no dose limiting toxicity (DLT) was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level.
- IPH2101 0.003 mg/kg: Participants were administered an IV dose of 0.003 mg/kg IPH2101 every 4 weeks for 4 cycles. Initially, 3 participants were treated at one dose level. If no dose limiting toxicity (DLT) was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level.
- IPH2101 0.015 mg/kg: Participants were administered an IV dose of 0.015 mg/kg IPH2101 every 4 weeks for 4 cycles. Initially, 3 participants were treated at one dose level. If no dose limiting toxicity (DLT) was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level.
- IPH2101 0.075 mg/kg: Participants were administered an IV dose of 0.075 mg/kg IPH2101 every 4 weeks for 4 cycles. Initially, 3 participants were treated at one dose level. If no dose limiting toxicity (DLT) was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level.
- IPH2101 0.3mg/kg: Participants were administered an IV dose of 0.3mg/kg IPH2101 every 4 weeks for 4 cycles. Initially, 3 participants were treated at one dose level. If no dose limiting toxicity (DLT) was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level.
- IPH2101 1mg/kg: Participants were administered an IV dose of 1 mg/kg IPH2101 every 4 weeks for 4 cycles. Initially, 3 participants were treated at one dose level. If no dose limiting toxicity (DLT) was observed, the dose was escalated to next higher level. If a DLT was observed among 1 of 3 treated participants in the first course at a dose level, 3 participants were additionally enrolled and treated at the same dose level. If no further DLT was observed during the first course in these additional participants, the dose was escalated to next higher dose level.
- IPH2101 3 mg/kg: Participants were administered an IV dose of 3mg/kg IPH2101 every 4 weeks for 4 cycles. Initially, 3 participants were treated at one dose level.If MTD this is not reached at 3mg/kg, 7 subjects will be enrolled at this dose to obtain more data from a larger subject pool to better evaluate safety, PK, PD and signs of efficacy.
Arm/Group | IPH2101 0.0003 mg/kg | IPH2101 0.003 mg/kg | IPH2101 0.015 mg/kg | IPH2101 0.075 mg/kg | IPH2101 0.3mg/kg | IPH2101 1mg/kg | IPH2101 3 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 3 | 10
Number of participants with DLT | 0 | 0 | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of IPH2101 After Cycle 1 Administration
Description: Cmax was obtained from the plasma concentration versus time data after IV administration of IPH2101.
Time Frame: Anti-KIR (1-7F9) concentrations were measured prior to infusion at 0.167, 1, 3, 6, 12 and 24 hours and then on Days 7, 14 and 21 after the start of the first dose administration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- IPH2101 0.0003 mg/kg; IPH2101 0.003 mg/kg; IPH2101 0.015 mg/kg: IV Bolus
- IPH2101 0.075 mg/kg; IPH2101 0.3 mg/kg; IPH2101 1 mg/kg; IPH2101 3 mg/kg: IV 1 hour infusion
Arm/Group | IPH2101 0.0003 mg/kg | IPH2101 0.003 mg/kg | IPH2101 0.015 mg/kg | IPH2101 0.075 mg/kg | IPH2101 0.3 mg/kg | IPH2101 1 mg/kg | IPH2101 3 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 6 | 3 | 3 | 10
ng/mL | 0 (0) | 45.8 (41.3) | 316 (53.8) | 1620 (38.4) | 4510 (30.9) | 24800 (25.5) | 55200 (31.7)

3. Secondary Outcome: Area Under the Plasma-concentration-time Curve [AUC (INF)] of IPH2101 After Cycle 1 Administration
Description: AUC(INF), area under the plasma concentration-time curve from zero to the last time of the last quantifiable concentration within the dosing interval was calculated for Cycle 1.
Time Frame: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hours/ml
Groups:
- IPH2101 0.0003 mg/kg; IPH2101 0.003 mg/kg; IPH2101 0.015 mg/kg: IV bolus injection
- IPH2101 0.3mg/kg; IPH2101 1 mg/kg; IPH2101 3 mg/kg: IV 1 hour infusion
Arm/Group | IPH2101 0.0003 mg/kg | IPH2101 0.003 mg/kg | IPH2101 0.015 mg/kg | IPH2101 0.075 mg/kg | IPH2101 0.3mg/kg | IPH2101 1 mg/kg | IPH2101 3 mg/kg
Number analyzed (Participants) | 2 | 3 | 3 | 5 | 2 | 3 | 10
ng*hours/ml | 0 (0) | 808 (49.7) | 16593 (273.3) | 161811 (61.5) | 596308 (0) | 4331537 (60.7) | 9292602 (41.7)

4. Secondary Outcome: Number of Evaluable Patients With Stable Disease. "Evaluable" is Defined as 2 Consecutive M Protein Assessments
Description: Disease Response Assessment by Principal Investigator and Sponsor(Efficacy Population).Stable Disease was defined as not meeting criteria for complete response, very good partial response, partial response, or progressive disease
Time Frame: From start of the treatment to end of study or disease progression
Measure: Number; unit: Number of participants
Groups:
- IPH2101 0.0003 mg/kg; IPH2101 0.003 mg/kg; IPH2101 0.015 mg/kg; IPH2101 0.075 mg/kg; IPH2101 0.3 mg/kg; IPH2101 1 mg/kg; IPH2101 3 mg/kg: Disease Response Assessment by Principal Investigator and Sponsor(Efficacy Population).Stable Disease was defined as not meeting criteria for complete response, very good partial response, partial response, or progressive disease
Arm/Group | IPH2101 0.0003 mg/kg | IPH2101 0.003 mg/kg | IPH2101 0.015 mg/kg | IPH2101 0.075 mg/kg | IPH2101 0.3 mg/kg | IPH2101 1 mg/kg | IPH2101 3 mg/kg
Number analyzed (Participants) | 1 | 2 | 2 | 5 | 0 | 3 | 6
Number of participants | 1 | 1 | 1 | 3 |  | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening and until the end of study at each study visit. Maximal study duration according to dose level was 4 to 9 months.
Description: All participants who received at least one dose of the study drug (safety population).
Arm/Group | 0.0003 mg/kg | 0.003 mg/kg | 0.015 mg/kg | 0.075 mg/kg | 0.3 mg/kg | 1 mg/kg | 3 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/3 | 5/6 | 0/3 | 0/3 | 3/10
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 6/6 | 3/3 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.0003 mg/kg (N=4) | 0.003 mg/kg (N=3) | 0.015 mg/kg (N=3) | 0.075 mg/kg (N=6) | 0.3 mg/kg (N=3) | 1 mg/kg (N=3) | 3 mg/kg (N=10)
Headeache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased platelets (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
progression of disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
worsening back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
worsening nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
infection with grade 4 neutrophil (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
elevated creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.0003 mg/kg (N=4) | 0.003 mg/kg (N=3) | 0.015 mg/kg (N=3) | 0.075 mg/kg (N=6) | 0.3 mg/kg (N=3) | 1 mg/kg (N=3) | 3 mg/kg (N=10)
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 4 (4)
chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Non Cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
edema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
blood creatinin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
white blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days